CLINICAL TRIAL: NCT05548712
Title: A Double-Blinded, Randomized-Control-Trial to Investigate the Effect of Pulsed Electromagnetic Field (PEMF) for Patients With Knee Osteoarthritis
Brief Title: The Effect of PEMF for Patients With Knee OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021.491
Record Dates: First submitted 2022-08-12; First posted 2022-09-21 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic
Keywords: Pulse electromagnetic field; PEMF; Knee Osteoarthritis; Knee OA; Knee pain
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into either treatment group or sham group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: It is doubled blinded, a subject 's specific ID card will be provided for each of the enrolled subject and the investigators don't know whether it is PEMF or Sham treatment for that subject's specific ID card. And the investigator will ask the manufactory about the number of grouping at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Device: Pulse Electromagnetic Field
- Sham group (Sham Comparator)
  Interventions: Device: Sham Pulse Electromagnetic Field

INTERVENTIONS:
Device: Pulse Electromagnetic Field — Subjects will receive PEMF treatment with the duration of 8 weeks, twice a week with total 16 treatment sessions and do the home-based exercise twice a week for 8 weeks.
  Arms: Treatment group
Device: Sham Pulse Electromagnetic Field — Subjects will receive sham PEMF treatment with the duration of 8 weeks, twice a week with total 16 treatment sessions and do the home-based exercise twice a week for 8 weeks.
  Arms: Sham group

SUMMARY:
Health care costs are increasing alarmingly, which will impose an overwhelming economic burden to an aging society like that of Hong Kong. For example, degenerative musculoskeletal disorders such as osteoarthritis (OA) present a grand challenge with its high prevalence (>40% in the elderly suffered from knee OA). OA is a debilitating progressive disease with typical symptoms such as acute pain causing loss of mobility Currently there is no cure for OA. Pharmacological treatment and new regenerative technologies such as stem cell therapy are actively being developed, but most of these options are very expensive per se, and side effects are not uncommon. Costeffectiveness is also a major consideration for devising new therapeutic modalities for OA.

There are emerging evidences showing that pulsed electromagnetic field (PEMF) can modulae mitochondrial activities for muscle gain. PEMF exposure on top of regular exercise training may promote muscle regeneration and tissue healing.

This study aims to conduct a double-blinded, randomized controlled trial to investigate the effect of PEMF treatment on knee pain in patients with knee OA. We hypothesize that PEMF treatment is effective to relief in pain and improve knee function in Knee OA subjects.

Based on the aim of this study, older adult patients (aged 50 or above) with knee OA with Kellgren-Lawrence grade 2-4 by X-ray, have sedentary lifestyle (Tegner activity level less or equal to 3), no acute knee injuries in past 12 months, no muscle strain in past 12 months and not degenerative joint disease in other joints except the involved knee.

To estimate the improvement of patients, isometric quadricep muscle strength, posture assessment, serum myokine level, serum vitamin D level and selfreported outcome with questionnaires will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 or above
2. knee OA with Kellgren-Lawrence grade 2-4 by X-ray
3. Sedentary lifestyle (Tegner activity level ≤ 3)
4. No acute knee injuries in past 12 months
5. No muscle strain in past 12 months
6. No degenerative joint diseases in other joints except the involved knee

Exclusion Criteria:

1. Age smaller than 50 years old
2. Experienced any concomitant bone fracture, ACL injury, major meniscus injury
3. Any rheumatological diseases
4. Metal implants that would cause interference on MRI
5. Previous contralateral knee injury
6. Recent knee injections (prior 3 months)
7. Physical inability to undertake testing procedures
8. Pregnancy or possibility of pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Change of Peak torque of Isometric muscle strength | pre PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF
  The peak torque in kgf will be recorded with in 2 trials in the 5 seconds isometric muscle strength test.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | pre PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF
  Consists of four items recording the subject's time of spending on physical activities during the past 7 days with a validated Chinese version of the quantitative physical activity questionnaire, and the physical activity level will be evaluated by Metabolic Equivalent of task(MET) per minute and classified as physical level with Low, Moderate or High.
Tegner activity score | pre PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF
  This is an activity level scaled from 1 (low activity) to 10 (high activity).
Short Form-36 questionnaires (SF-36) | pre PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF
  This is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Serum myokine evaluation | pre PEMF treatment, 3-months, 6-months, and 12-months after the commencement of PEMF
  Phlebotomy (5ml) will be performed on the day before PEMF treatment, at 4- and 8- weeks after commencement of treatment, and at 8 months after the commencement of intervention. The serum will be prepared by centrifugation and kept in a -80o freezer until use. Quantitative analysis for myokines and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme-linked immunosorbent assay (ELISA) and report with pg/ml. These include Brain-derived neurotrophic factor (BDNF), Fibroblast growth factor-21 (FGF-21), Interleukin-6 (IL-6), IL-15, Irisin, Myostatin (MSTN)/GDF8, Insulin-like growth factor 1 (IGF-1), FGF-2, IL-8, Follistatin, Musclin, Myonectin, Decorin, Meteorinlike, Osteopontin, Secreted protein acidic and rich in cysteine (SPARC), Klotho, Procollagen type III Nterminal peptide (P3NP), and C- terminal of troponin T1 (TNNT1).
The speed and rate of force development in 6 repetitions in chair stand test | pre PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF
  The rate of force development will be determined as the mean slope of the rising force of the first force peak of each of the 2nd to the 6th repetition in the interval of 30-70% exerted peak force. Results are reported as the mean of the two fastest approved trials in body weight per second (BW/s).
Change of centre of pressure with the position of double leg squat | pre PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF
  The centre of pressure excursion range in the anterior-posterior direction in mm will be recored.
Change of centre of pressure with the position of static postural codition | pre PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF
  The centre of pressure excursion range in the anterior-posterior direction in mm will be recored.
Change of centre of pressure with the position of dynamic postural codition | pre PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF
  The centre of pressure excursion range in the anterior-posterior direction in mm will be recored.
Serum vitamin D level and vitamin D metabolites evaluation | pre PEMF treatment, 3-months, 6-months, and 12-months after the commencement of PEMF
  Blood samples will be taken under non-fasting conditions. Serum / plasma obtained will be immediately stored at -80°C until analysis. Serum 25(OH) Vit-D assay: Serum 25(OH)Vit-D levels will be measured by commercial 25(OH) Vitamin D ELISA kit (Abcam ab213966) according to the manufacturer's instruction, providing the quantitative determination of 25(OH) Vitamin D3 and 25(OH) Vitamin D2. Sensitivity: 1.98 ng/ml (Range: 0.5 ng/ml - 1010 ng/ml).
Visual Analogue Scale | pre PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF
  The subjective measurement for chronic and acute pain will be recorded by the Visual Analogue Scale (VAS). VAS consists of a 10-cm line which represents the continuum between "painless" and "worst pain from 0 cm to 10 cm. The subject will be asked to draw a mark of it before and after each PEMF treatment session.
Change of the scoring of Knee injury and Osteoarthritis Outcome Score | pre PEMF treatment , 2-months, 3-months, 6-months, and 12-months after the commencement of PEMF
  Consist of 42 items with 5 subscapes: pain, other symptoms, function in daily living (ADL), function in sport and recreation (Sport/Rec), and knee-related quality of life (QOL) from 0% to 100% where higher score indicate a better outcome in each subscape.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tim-Yun Ong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewers

DOCUMENTS (2):
  • Study Protocol (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT05548712/Prot_000.pdf
  • Informed Consent Form (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT05548712/ICF_001.pdf